CLINICAL TRIAL: NCT01884753
Title: Correlations of 3D Urethral and Paraurethral Sonographic Findings With Urodynamic Studies, Lower Urinary Tract Symptoms & Sexual Dysfunction in Female Patients With Lower Urinary Tract Symptoms.
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 102021-F
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2021-08

CONDITIONS: Lower Urinary Tract Dysfunction; Overactive Bladder Syndrome
Keywords: lower urinary tract symptoms; overactive bladder syndrome; antimuscarinic drug; three-dimensional power Doppler ultrasound; sexual dysfunction
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult women with lower urinary tract symptoms: Adult women (not less than 20 year-old) with lower urinary tract symptoms

SUMMARY:
The main purpose of this study is to get the urethra and pelvic sonographic imaging by 4D ultrasound examinations, and to correlate the sonographic findings with urodynamic variables, pad weights and LUTS. Besides, the associations of the blood flow of vagina/urethra and sexual dysfunction can be explored.

DETAILED DESCRIPTION:
Female lower urinary tract dysfunction includes stress urinary incontinence, overactive bladder syndrome and voiding dysfunction. There are a lot of bladder studies, such as researches of bladder wall thickness and bladder volume. However, there were few studies of urethra for female patients with lower urinary tract symptoms (LUTS), especially for storage disorder. Thus, the main purpose of this study is to get the urethra and pelvic sonographic imaging by 4D ultrasound examinations, and to correlate the sonographic findings with urodynamic variables, pad weights and LUTS. The investigators hope to identify important LUTS sonographic biomarkers that can be used by primary physicians as a tool for assess female LUTS, and thus decreasing the need of further invasive urodynamic studies.

Besides, the associations of the blood flow of vagina/urethra and sexual dysfunction (assessed by female sexual function index) can be explored.

In addition, women who receive antimuscarinics treatment will receive follow-up 4D imaging and request to complete questionnaire 12 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Women with lower urinary tract symptoms
* Not less than 20 years-old

Exclusion Criteria:

* Patients with a history of stroke.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with lower urinary tract symptoms
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2014-02-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Urethral/pelvic blood flow perfusion pattern between subgroups of women with lower urinary tracts | 1 day
  We will get the associations of urethral/pelvic blood flow perfusion pattern between subgroups of women with lower urinary tracts, and the above results will be compared to that of the asymptomatic control group.

SECONDARY OUTCOMES:
Urethral/pelvic blood flow perfusion pattern after antimuscarinics | 12 weeeks
  We will compare the urethral/pelvic blood flow perfusion pattern between the baseline and 12 weeks' antimuscarinic treatment (solifenacin 5 mg SR qd or tolerodine 4 mg ER qd) in women with overactive bladder syndrome.

OTHER OUTCOMES:
The subgroup differences of urethral/pelvic volume, hiatal area and rupture of puborectalis muscles | 1 day
  we will use 4 D ultrasound to assess the urethral/pelvic volume, hiatal area and rupture of puborectalis muscles among subgroups of women with lower urinary tract symptoms, and the above results will be compared to that of the control group. Besides, the correlation of imaging findings and clinical symptoms (such as lower urinary tract symptoms and sexual dysfunction) will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Mou Hsiao, MD, Principal Investigator — Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan